CLINICAL TRIAL: NCT01694758
Title: OPtimal Type 2 dIabetes Management Including Benchmarking and Standard Treatment in CEEMEA (OPTIMISE)
Brief Title: OPtimal Type 2 dIabetes Management Including Benchmarking and Standard Treatment in CEEMEA
Acronym: OPTIMISE
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CME-XXX-2012/1
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
Keywords: Benchmarking could improve quality of patient care; ESC and ATP III Guidelines
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with diabetes type 2

SUMMARY:
OPTIMISE-CEEMEA is a multinational, multi-centre, observational, prospective study which will include patients suffering from diabetes type 2, treated or untreated, insulin dependent or not insulin dependent.

In this study we aim to explore at a primary care level whether the use of benchmarking against a set of guideline-based reference values on a patient basis, may improve quality of patient care, in particular control of diabetes, lipids and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from diabetes type 2,
* treated or untreated,
* insulin dependent or not insulin dependent Able to read and send SMS (if SMS applicable)

Exclusion Criteria:

* Type 1 diabetes Pregnancy diabetes
* Hospitalization at the moment of enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes type 2
Sampling Method: Non-Probability Sample
Enrollment: 733 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in the benchmarking group achieving pre-set targets for HbA1c1 | after 12 months of follow-up
  To investigate whether the use of benchmarking could improve quality of patient care, in particular the control of diabetes, lipids and blood pressure, expressed as the percentage of patients in the benchmarking group achieving pre-set targets for HbA1c1

SECONDARY OUTCOMES:
Quality of patient care improvement, in particular the control of diabetes, lipids and blood pressure | after 12 months of follow-up versus baseline
  To investigate whether the use of benchmarking could improve quality of patient care, in particular the control of diabetes, lipids and blood pressure
Markers of preventive screening | after 12 months of follow-up versus baseline
  To follow up evolution markers of preventive screening; retinopathy, neuropathy, dietary counseling, smoking habits, BMI, waist circumference, physical activity
The LDL cholesterol parameter of the primary and secondary objectives according to ATP III guidelines | after 12 months of follow-up versus baseline
  To investigate the LDL cholesterol parameter of the primary and secondary objectives according to ATP III guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Dan Isacoff, ASSOC. PROF., Principal Investigator — University of Medicine and Pharmacy Carol Davila, Bucharest, Romania
Locations (20):
- Bulgaria (4):
  - Research Site, Blagoevgrad
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sofia
- Romania (16):
  - Research Site, Alexandria
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Constanța
  - Research Site, Craiova
  - Research Site, Galati
  - Research Site, Giurgiu
  - Research Site, Iași
  - Research Site, Oradea
  - Research Site, Piteşti
  - Research Site, Ploieşti
  - Research Site, Satu Mare
  - Research Site, Tg Jiu
  - Research Site, Tg Mures
  - Research Site, Timișoara